CLINICAL TRIAL: NCT00226915
Title: Randomized Phase III Trial of Conventional Paclitaxel and Carboplatin Versus Dose Dense Weekly Paclitaxel and Carboplatin in Patients With Newly Diagnosed Stage II-IV Mullerian Carcinoma
Brief Title: Trial of Tri-weekly TJ Versus Weekly TJ for Stage II-IV Mullerian Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japanese Gynecologic Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JGOG3016; C000000183 (by UMIN)
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Epithelial Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
Keywords: ovarian neoplasms; randomized controlled trial; paclitaxel; carboplatin
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Drug: Paclitaxel 180mg/m2＋CBDCA AUC6 q21 days x 6-9cycles
  Interventions: Drug: Paclitaxel+Carboplatin
- 2 (Experimental): Drug: Paclitaxel 80mg/m2 weekly ＋CBDCA AUC6 q21 days x 6-9cycles
  Interventions: Drug: Paclitaxel+Carboplatin

INTERVENTIONS:
Drug: Paclitaxel+Carboplatin — Paclitaxel 180mg/m2＋CBDCA AUC6 q21 days x 6-9cycles
  Arms: 1
Drug: Paclitaxel+Carboplatin — Paclitaxel 80mg/m2 weekly ＋CBDCA AUC6 q21 days x 6-9cycles
  Arms: 2

SUMMARY:
The purpose of the study is to compare progression-free survival of conventional paclitaxel and carboplatin vs weekly paclitaxel and carboplatin in patients with newly diagnosed stage II-IV ovarian epithelial, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
This is a randomized, multicenter study. Patients are stratified according to residual disease 1 cm or less vs more than 1cm, stage II vs III vs IV, and histology (clear cell or mucinous vs. serous or others). Patients are randomized to one of two treatment arms.

Arm I: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 60 minutes on day 1 for 6-9 cycles.

Arm II: Patients receive paclitaxel IV over 1 hour days 1, 8, and 15 and carboplatin IV over 60 minutes on day 1 for 6-9 cycles.

In both arms, cycles repeat 6 cycles every 21 days in the absence of disease progression or unacceptable toxicity. Additional 3 cycles are given if clinical partial or complete response after 6 cycles.

PROJECTED ACCRUAL: A total 600 patients (300 per treatment arm) will be accrued for this study within 3 years. Assuming median progression-free survivals of 16 months and 21 months and a recruitment period of 3 years this can be achieved by recruiting 600 patients designed to have 80 % detect to a difference between the two arms at the two-sided 5% level of statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage II-IV ovarian epithelial, primary peritoneal, or fallopian tube cancer
* No prior chemotherapy
* Age: 20 and more
* Performance status: ECOG 0-3
* 1) Absolute neutrophil count at least 1,500/mm3 2) Platelet count at least 100,000/mm3 3) Bilirubin less than 1.5mg/dL 4) SGOT less than 100 IU/l 5) Serum creatinine less than 1.5mg/dL
* Written informed consent

Exclusion Criteria:

* Patients with ovarian borderline tumor
* Patients who have any evidence of the other cancer present within the last 5 years with the exception of carcinoma in situ or intramucosal cancer that is curable with local therapy
* Patients with active infection or uncontrolled diabetes
* Patients with unstable angina, or those who have had a myocardial infarction within the past 6 months, or patients with serious arrythmia that requires medication
* Patients who have a history of hypersensitivity to polyoxyethylated castor oil (Cremophor EL)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2003-04 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Suvaival | During the protocol treatment then 18 months from the last day of the protocol treatment
  From the registration date, the earliest observed event from any of the following events 1. Death from any cause death date 2. The date of the first diagnostic imaging examination that confirmed exacerbation and recurrence.
  Clinical exacerbation diagnosis date if not based on diagnostic imaging 3. If none of the above events are observed, the most recent outpatient consultation date / in hospital

SECONDARY OUTCOMES:
Overall Survival | During the protocol treatment then 18 months from the last day of the protocol treatment
  The period from the registration date to the date of death due to any cause. In the case of survivors, the final surviving confirmation date will be censored.
  In the case of untraceable cases, the last surviving confirmation date before tracking becomes impossible will be censored.
QOL | During the protocol treatment then 18 months
  QOL assessed by FACT-Taxane(Version 4A)
Adverse Event | During the protocol treatment then 18 months
  Adverse Event assessed by CTC(Version 2.0 Japanese version)

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Yasuda, M.D., Study Chair — The Jikei University School of Medicine
Locations (1):
- National Cancer Center Hospital, Chuo-ku, Tokyo, Japan

REFERENCES:
- [Background] McGuire WP, Hoskins WJ, Brady MF, Kucera PR, Partridge EE, Look KY, Clarke-Pearson DL, Davidson M. Cyclophosphamide and cisplatin compared with paclitaxel and cisplatin in patients with stage III and stage IV ovarian cancer. N Engl J Med. 1996 Jan 4;334(1):1-6. doi: 10.1056/NEJM199601043340101. PMID 7494563
- [Background] Citron ML, Berry DA, Cirrincione C, Hudis C, Winer EP, Gradishar WJ, Davidson NE, Martino S, Livingston R, Ingle JN, Perez EA, Carpenter J, Hurd D, Holland JF, Smith BL, Sartor CI, Leung EH, Abrams J, Schilsky RL, Muss HB, Norton L. Randomized trial of dose-dense versus conventionally scheduled and sequential versus concurrent combination chemotherapy as postoperative adjuvant treatment of node-positive primary breast cancer: first report of Intergroup Trial C9741/Cancer and Leukemia Group B Trial 9741. J Clin Oncol. 2003 Apr 15;21(8):1431-9. doi: 10.1200/JCO.2003.09.081. Epub 2003 Feb 13. PMID 12668651
- [Background] Heintz AP, Odicino F, Maisonneuve P, Beller U, Benedet JL, Creasman WT, Ngan HY, Sideri M, Pecorelli S. Carcinoma of the ovary. J Epidemiol Biostat. 2001;6(1):107-38. No abstract available. PMID 11385772
- [Background] Strnad CM, Grosh WW, Baxter J, Burnett LS, Jones HW 3rd, Greco FA, Hainsworth JD. Peritoneal carcinomatosis of unknown primary site in women. A distinctive subset of adenocarcinoma. Ann Intern Med. 1989 Aug 1;111(3):213-7. doi: 10.7326/0003-4819-111-3-213. PMID 2502058
- [Background] Feuer GA, Shevchuk M, Calanog A. Normal-sized ovary carcinoma syndrome. Obstet Gynecol. 1989 May;73(5 Pt 1):786-92. PMID 2704507
- [Background] Piccart MJ, Bertelsen K, James K, Cassidy J, Mangioni C, Simonsen E, Stuart G, Kaye S, Vergote I, Blom R, Grimshaw R, Atkinson RJ, Swenerton KD, Trope C, Nardi M, Kaern J, Tumolo S, Timmers P, Roy JA, Lhoas F, Lindvall B, Bacon M, Birt A, Andersen JE, Zee B, Paul J, Baron B, Pecorelli S. Randomized intergroup trial of cisplatin-paclitaxel versus cisplatin-cyclophosphamide in women with advanced epithelial ovarian cancer: three-year results. J Natl Cancer Inst. 2000 May 3;92(9):699-708. doi: 10.1093/jnci/92.9.699. PMID 10793106
- [Background] Muggia FM, Braly PS, Brady MF, Sutton G, Niemann TH, Lentz SL, Alvarez RD, Kucera PR, Small JM. Phase III randomized study of cisplatin versus paclitaxel versus cisplatin and paclitaxel in patients with suboptimal stage III or IV ovarian cancer: a gynecologic oncology group study. J Clin Oncol. 2000 Jan;18(1):106-15. doi: 10.1200/JCO.2000.18.1.106. PMID 10623700
- [Background] International Collaborative Ovarian Neoplasm Group. Paclitaxel plus carboplatin versus standard chemotherapy with either single-agent carboplatin or cyclophosphamide, doxorubicin, and cisplatin in women with ovarian cancer: the ICON3 randomised trial. Lancet. 2002 Aug 17;360(9332):505-15. doi: 10.1016/S0140-6736(02)09738-6. PMID 12241653
- [Background] Alberts DS, Green S, Hannigan EV, O'Toole R, Stock-Novack D, Anderson P, Surwit EA, Malvlya VK, Nahhas WA, Jolles CJ. Improved therapeutic index of carboplatin plus cyclophosphamide versus cisplatin plus cyclophosphamide: final report by the Southwest Oncology Group of a phase III randomized trial in stages III and IV ovarian cancer. J Clin Oncol. 1992 May;10(5):706-17. doi: 10.1200/JCO.1992.10.5.706. PMID 1569443
- [Background] Eisenhauer EA, ten Bokkel Huinink WW, Swenerton KD, Gianni L, Myles J, van der Burg ME, Kerr I, Vermorken JB, Buser K, Colombo N, et al. European-Canadian randomized trial of paclitaxel in relapsed ovarian cancer: high-dose versus low-dose and long versus short infusion. J Clin Oncol. 1994 Dec;12(12):2654-66. doi: 10.1200/JCO.1994.12.12.2654. PMID 7989941
- [Background] Bois AD, Lueck HJ, Meier W, Moebus V, Costa SD, Bauknecht T, Richter B, Warm M, Schroeder W, Olbricht S, Nitz U, Jackisch C. Cisplatin/Paclitaxel Vs Carboplatin/Paclitaxel in Ovarian Cancer: Update of an Arbeitsgemeinschaft Gynaekologische Onkologie (AGO) Study Group Trial. American Society of Clinical Oncology 18:356a(Abstract 1374), 1999.
- [Background] Ozols R, Bundy B, Fowler J, Clarke-Pearson D, Mannel R, Hartenbach E , Baergen R. Randomized Phase III Study of Cisplatin (CIS)/Paclitaxel (PAC) Versus Carboplatin (CARBO)/PAC in Optimal Stage III Epithelial Ovarian Cancer (OC): A Gynecologic Oncology Group Trial (GOG 158). American Society of Clinical Oncology 18:356a(Abstract.1373), 1999.
- [Background] Bertelsen K, Jakobsen A, Stroyer J, Nielsen K, Sandberg E, Andersen JE, Ahrons S, Nyland M, Hjortkjaer Pedersen P, Larsen G, et al. A prospective randomized comparison of 6 and 12 cycles of cyclophosphamide, adriamycin, and cisplatin in advanced epithelial ovarian cancer: a Danish Ovarian Study Group trial (DACOVA). Gynecol Oncol. 1993 Apr;49(1):30-6. doi: 10.1006/gyno.1993.1081. PMID 8482557
- [Background] Hakes TB, Chalas E, Hoskins WJ, Jones WB, Markman M, Rubin SC, Chapman D, Almadrones L, Lewis JL Jr. Randomized prospective trial of 5 versus 10 cycles of cyclophosphamide, doxorubicin, and cisplatin in advanced ovarian carcinoma. Gynecol Oncol. 1992 Jun;45(3):284-9. doi: 10.1016/0090-8258(92)90305-3. PMID 1612505
- [Background] Planner RS, Allen DG, Brand AH, Grant PT, Toner GC, Sykes PH. Paclitaxel (Taxol) as salvage therapy for relapsed ovarian cancer. Aust N Z J Obstet Gynaecol. 1996 May;36(2):168-70. doi: 10.1111/j.1479-828x.1996.tb03278.x. PMID 8798307
- [Background] Hudis C. New approaches to adjuvant chemotherapy for breast cancer. Pharmacotherapy. 1996 May-Jun;16(3 Pt 2):88S-93S. PMID 8726587
- [Background] Tan G, Heqing L, Jiangbo C, Ming J, Yanhong M, Xianghe L, Hong S, Li G. Apoptosis induced by low-dose paclitaxel is associated with p53 upregulation in nasopharyngeal carcinoma cells. Int J Cancer. 2002 Jan 10;97(2):168-72. doi: 10.1002/ijc.1591. PMID 11774260
- [Background] Torres K, Horwitz SB. Mechanisms of Taxol-induced cell death are concentration dependent. Cancer Res. 1998 Aug 15;58(16):3620-6. PMID 9721870
- [Background] Fennelly D, Aghajanian C, Shapiro F, O'Flaherty C, McKenzie M, O'Connor C, Tong W, Norton L, Spriggs D. Phase I and pharmacologic study of paclitaxel administered weekly in patients with relapsed ovarian cancer. J Clin Oncol. 1997 Jan;15(1):187-92. doi: 10.1200/JCO.1997.15.1.187. PMID 8996141
- [Background] Bremer K. Weekly Paclitaxel/Carboplatin as First-Line Chemotherapy in Advanced Ovarian Cancer. American Society of Clinical Oncology 18:367a(Abstract. 1419), 1999.
- [Background] Katsumata N, Watanabe T, Mukai H, Kasamatsu T, Tsunematsu R, Yamada T, Ohmi K. A Phase II Trial of Weekly Paclitaxel/Carboplatin (TJ) as Salvage Chemotherapy in Patients with Relapsed Ovarian Cancer. American Society of Clinical Oncology 20:217a(Abstract. 865), 2001.
- [Background] Belani C, Barstis J, Perry M, Larocca R, Nattam S, Clark R, Rinaldi D, Mills G. Phase II Multicenter Randomized Trial of Weekly Paclitaxel (P) Administered in Combination with Carboplatin (C) Followed by Maintenance P Vs. Observation for Patients (Pts.) with Advanced & Metastatic Non-Small Cell Lung Cancer (NSCLC). American Society of Clinical Oncology 20:323a(Abstract. 1287), 2001.
- [Background] Yasuda M, Kimura E, Ochiai K, Tada S, Udagawa Y, Aoki D, Nozawa S, Kikuchi Y, Kita T, Nishida M, Tsunoda H. [Dose finding study of paclitaxel and carboplatin for ovarian cancer (JKTB)]. Gan To Kagaku Ryoho. 2001 Apr;28(4):493-8. Japanese. PMID 11329783
- [Background] Onnis A, Marchetti M, Padovan P, Castellan L. Neoadjuvant chemotherapy in advanced ovarian cancer. Eur J Gynaecol Oncol. 1996;17(5):393-6. PMID 8933839
- [Background] Aure JC, Hoeg K, Kolstad P. Clinical and histologic studies of ovarian carcinoma. Long-term follow-up of 990 cases. Obstet Gynecol. 1971 Jan;37(1):1-9. No abstract available. PMID 4321469
- [Background] Bois A, Weber B, Pfisterer J, Goupil A, Wagner U, Barats J, Olbricht S, Mousseau M, Nitz U, Meden H. Epirubicin/Paclitaxel/Carboplatin (TEC) Vs. Paclitaxel/Carboplatin (TC) in First-Line Treatment of Ovarian Cancer FIGO Stages IIb-IV. Interim Results of an AGO-GINECO Intergroup Phase III Trial. American Society of Clinical Oncology 20:202a(Abstract.805), 2001.
- [Derived] Harano K, Terauchi F, Katsumata N, Takahashi F, Yasuda M, Takakura S, Takano M, Yamamoto Y, Sugiyama T. Quality-of-life outcomes from a randomized phase III trial of dose-dense weekly paclitaxel and carboplatin compared with conventional paclitaxel and carboplatin as a first-line treatment for stage II-IV ovarian cancer: Japanese Gynecologic Oncology Group Trial (JGOG3016). Ann Oncol. 2014 Jan;25(1):251-7. doi: 10.1093/annonc/mdt527. PMID 24356636
- [Derived] Katsumata N, Yasuda M, Isonishi S, Takahashi F, Michimae H, Kimura E, Aoki D, Jobo T, Kodama S, Terauchi F, Sugiyama T, Ochiai K; Japanese Gynecologic Oncology Group. Long-term results of dose-dense paclitaxel and carboplatin versus conventional paclitaxel and carboplatin for treatment of advanced epithelial ovarian, fallopian tube, or primary peritoneal cancer (JGOG 3016): a randomised, controlled, open-label trial. Lancet Oncol. 2013 Sep;14(10):1020-6. doi: 10.1016/S1470-2045(13)70363-2. Epub 2013 Aug 13. PMID 23948349
- [Derived] Katsumata N, Yasuda M, Takahashi F, Isonishi S, Jobo T, Aoki D, Tsuda H, Sugiyama T, Kodama S, Kimura E, Ochiai K, Noda K; Japanese Gynecologic Oncology Group. Dose-dense paclitaxel once a week in combination with carboplatin every 3 weeks for advanced ovarian cancer: a phase 3, open-label, randomised controlled trial. Lancet. 2009 Oct 17;374(9698):1331-8. doi: 10.1016/S0140-6736(09)61157-0. Epub 2009 Sep 18. PMID 19767092
- See also: Please refer "ongoing studies" (in Japanese) — http://www.jgog.gr.jp/